CLINICAL TRIAL: NCT06947044
Title: Biomarkers in Patients With Anemia-Induced Thrombocytopenic Bleeding (BAIT): A Pilot Study
Brief Title: Biomarkers in Patients With Anemia-Induced Thrombocytopenic Bleeding
Acronym: BAIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donald Arnold (Other)
Responsible Party: Sponsor-Investigator, Donald Arnold, Principal Investigator, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15529
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Leukemia; Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukaemia
Keywords: transfusion; red blood cells; hemoglobin level; bleeding
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RBC transfusion strategy to maintain a hemoglobin level of at least 110 g/LL (Experimental): Participants randomized to this arm will be assigned to a liberal RBC transfusion strategy to maintain a hemoglobin level of at least 110 g/L.
  Interventions: Procedure: RBC transfusion strategy
- Standard-of-care RBC transfusion strategy (No Intervention): Participants randomized to this arm will be assigned to a restrictive RBC transfusion strategy of standard-of-care, which is typically to maintain a hemoglobin level of at least 70-80 g/L.

INTERVENTIONS:
Procedure: RBC transfusion strategy — RBC transfusion strategy to maintain a hemoglobin level of at least 110 g/L.
  Arms: RBC transfusion strategy to maintain a hemoglobin level of at least 110 g/LL

SUMMARY:
This pilot study aims to gather preliminary evidence on how different hemoglobin levels impact blood biomarkers related to bleeding. The feasibility of conducting a future larger clinical trial will also be assessed. Red blood cell transfusions are part of the standard of care for patients with leukemia. This study evaluates two transfusion strategies: one that maintains hemoglobin levels above the standard-of-care threshold, reflecting current routine practice; and another that maintains hemoglobin levels above 110 g/L, which is closer to the normal hemoglobin range. The normal hemoglobin range is 120-160 g/L for females and 140-180 g/L for males. Raising hemoglobin levels closer to normal values may reduce bleeding risk.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Inpatient
3. Diagnosis of acute myeloid leukemia or acute lymphocytic leukemia.
4. Less than 5 days have elapsed since the start of induction chemotherapy treatment.
5. Hemoglobin at enrolment is under 130 g/L.

Exclusion Criteria:

1. Failure to provide informed consent.
2. Unwilling to receive blood transfusions.
3. Life expectancy <72 hours.
4. Undergoing palliative chemotherapy.
5. Requires specialized blood products (e.g., antigen-matched, irradiation, etc.).
6. Diagnosis of acute promyelocytic leukemia.
7. Diagnosis of hyperleukocytosis (a white blood cell count exceeding 100 × 10^9/L).
8. Diagnosed with coagulopathies or ongoing treatment with therapeutic anticoagulants, aspirin or nonsteroidal anti-inflammatory drugs (history of inherited or acquired coagulation disorder, known hemolytic disease, INR > 1.5)
9. Evidence of iron overload (ferritin >800 ng/mL, transferrin saturation >80%) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Effect of maintaining a higher hemoglobin level (110 g/L) compared with the standard hemoglobin level on bleeding-related biomarkers. | Samples will be collected before chemotherapy onset, and on days 7, 14, and 28. The first day of chemotherapy is considered day 1
  Blood and urine samples will be taken from participants at selected timepoints to measure levels of biomarkers from the endothelial integrity, inflammation, and fibrinolysis/coagulation domains.
Protocol adherence to the study intervention (feasibility outcome) | Day 1 to 30
  The total number of days where hemoglobin levels were above the assigned threshold or days where RBCs were administered when the hemoglobin level was reported to be below that threshold.
Protocol adherence to the study schedule (feasibility outcome) | Day 1 to 30
  Measurement of how consistently participants and study staff follow the prescribed schedule for study assessments and sample collections as outlined in the study protocol. Measurements include percentage of scheduled biomarker testing days with data collected, percentage of non-weekday study days with completed bleeding assessments, and percentage of scheduled study days with completed FACT questionnaires.
Consent rate (feasibility outcome) | Through study completion, an average of 1.5 years
  The proportion of potential participants who agree to participate in the study.
Screen failure rate (feasibility outcome) | Through study completion, an average of 1.5 years
  The proportion of participants who are screened for eligibility but do not meet the study's inclusion and exclusion criteria and are therefore not enrolled in the trial.

SECONDARY OUTCOMES:
The total number of blood products administered to participants in the liberal and standard arms of the study | Day 1 to 30
  The number of platelet and red blood cell units administered to each participant will be summed and compared between study groups.
The association between the hemoglobin threshold used and bleeding events | Day 1 to 30
  Comparison of the time-to-bleed data between the study groups.
The association between the hemoglobin threshold used and quality-of-life | Assessed weekly, from before chemotherapy onset to day 28
  The FACIT-Thrombocytopenia scale will be used to score participants between 0 (worst quality of life) and 52 (best quality of life). Higher scores indicate better quality of life, and less impact of symptoms related to thrombocytopenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided